CLINICAL TRIAL: NCT04435418
Title: Eliquis Acute Stroke Safety Evaluation
Acronym: EASSE
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Ken Butcher, Professor, University of Alberta
Other Study IDs: Version 1.0 September 30, 2016
Record Dates: First submitted 2020-06-14; First posted 2020-06-17 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack; Atrial Fibrillation
Keywords: Atrial fibrillation; Ischemic stroke; Hemorrhagic transformation; Apixaban; Cardioembolic stroke; Intracerebral hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Atrial Fibrillation; Embolic Stroke; Cerebral Hemorrhage | interventions — apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Apixaban — The decision to treat with apixaban and the timing of initiation will be at the attending physicians' discretion, independent of enrolment in EASSE.
  Other Names: Eliquis

SUMMARY:
Study Design:

This is an investigator-initiated prospective, open label, single arm phase IV study. Patients with documented non-valvular atrial fibrillation (AF) with acute TIA (defined as acute focal neurological deficits, with complete resolution of symptoms within 24 h of onset) or ischemic stroke, irrespective of infarct volume or clinical severity will be enrolled.

Study Aim and Objectives:

The overall aim of this study is to demonstrate the feasibility and safety of initiating apixaban therapy within 14 days of TIA or ischemic stroke regardless of the size and severity in patients with AF. Investigators will systematically assess prospectively collected CT scan images for evidence of HT and re-infarction.

DETAILED DESCRIPTION:
Study Hypothesis:

Investigators hypothesize that early initiation of apixaban within the first 14 days of stroke or TIA is not associated with increased symptomatic intracranial haemorrhage.

Study Design:

EASSE is an investigator-initiated prospective, open label, single arm phase IV study. Consecutive patients with AF (new onset or previous history) with acute ischemic stroke or TIA will be screened from Emergency Department or stroke unit. A total of 100 patients will be recruited within 24 hours of initiation of apixaban after TIA or stroke. All study participants will be followed for 90 days after apixaban initiation. A National Institute of Health Stroke Scale (NIHSS) score, modified Rankin Scale (mRS), and Montreal Cognitive Assessment (MoCA) will be collected at baseline, 7, and 90 days after enrolment. All patients will have a non-contrast CT scan at baseline (within 24 hours from study recruitment) and at 7±2 days after enrolment. In the event of clinical deterioration, a repeat CT scan will be performed immediately.

Administrative Structure:

Case report forms and data monitoring will be completed on site. All imaging data will be read centrally at the Stroke Imaging Laboratory at the University of Alberta.

Procedures:

Apixaban therapy: The apixaban dose will be determined by the treating physician, based on age, weight and renal function as per the product monograph. Patients with two of the following: Age > 80, weight < 60 kg, and creatinine ≥ 133 (1.5 mg/dl), will have received 2.5 mg twice a day. All other patients will have received 5 mg twice a day.

Imaging Procedures and Analysis:

Anonymized dicom CT data will be analyzed centrally. Baseline infarct volumes will be measured using planimetric techniques and recurrent infarctions will be identified. Any HT seen at baseline and day 7 will be graded using European Cooperative Acute Stroke Study (ECASS) criteria.

Endpoints:

The primary endpoint is the symptomatic HT, defined as PH2 associated with a ≥4-point increase in NIHSS score within 90 days of initiating apixaban therapy. Secondary outcomes include any HT at day 7, systemic hemorrhagic complications, and recurrent ischemic events within 90 days of enrolment. Investigators will report serious adverse events (SAE) within the study period using standardized event, resolution and association codes, and they will be reported to the local Human Research Ethics Board.

Sample Size:

A sample of 100 patients is planned in order to obtain estimates of the frequency of symptomatic and asymptomatic HT associated with early apixaban initiation. The maximum acceptable rate of symptomatic HT is considered 2%, based on a meta-analysis of low molecular weight heparin treatment in acute stroke, indicating the absolute symptomatic HT rate ranged from 2.4% to 2.9%.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients
2. Must be ≥ 18 years of age.
3. Diagnosis of ischemic stroke, or Transient Ischemic Attack (TIA, defined as acute focal neurological deficits, with complete resolution of symptoms within 24 h of onset). In cases where onset time cannot be established, it will be considered to be the time when patient was last known to be well.
4. CT scan or MRI, with findings consistent with an ischemic etiology of symptoms.
5. Atrial Fibrillation (AF, paroxysmal or persistent), confirmed with ECG/Holter monitor, or by history (clinical documentation of previous AF must be provided).
6. Patients prescribed apixaban by their treating physician following their stroke/TIA.
7. Ability to obtain consent from patient or legally authorized representative.

Exclusion Criteria:

1. Acute or chronic renal failure, defined as eGFR <30 ml/min (Cockcroft Gault formula).
2. Known hypersensitivity to apixaban.
3. Prior treatment with apixaban or any other novel oral anticoagulant (including all Factor Xa antagonists). Treatment with warfarin prior to the stroke/TIA is acceptable, but enrolment cannot begin until the INR is ≤2.0.
4. Any significant ongoing systemic bleeding risk, i.e. active GI/GU bleeding or recent major surgery.
5. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
6. Recent past history or clinical presentation of ICH, subarachnoid haemorrhage (SAH), arterio-venous (AV) malformation, aneurysm, or cerebral neoplasm.
7. Hereditary or acquired haemorrhagic diathesis.
8. Stroke mimics (such as seizures, migraine etc.)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke (regardless of the size and severity ) or TIA in patients ≥ 18 years of age, with atrial fibrillation (newly or previously diagnosed), who can be treated with apixaban following stroke.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
symptomatic HT | 90 days
  Defined as PH2 associated with a ≥4-point increase in NIHSS score within 90 days of initiating apixaban therapy

SECONDARY OUTCOMES:
HT | Day 7
  Symptomatic or asymptomatic
Systemic hemorrhagic complications | 90 days
  Systemic bleeding
Recurrent ischemic events | 90 days
  TIA, ischemic stroke, or systemic emboli

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

DOCUMENTS (1):
  • Study Protocol (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT04435418/Prot_000.pdf